CLINICAL TRIAL: NCT03614377
Title: Prospective Multicenter Observation Study on the Association Between the Severity of Device-detected Sleep-disordered Breathing and the Risk of Cardiac Arrhythmic Events
Brief Title: DEvice-Detected CArdiac Tachyarrhythmic Events and Sleep-disordered Breathing (DEDiCATES)
Acronym: DEDiCATES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: SMC 2017-03-017-010
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Sleep Disorder; Cardiac Arrythmias; Cardiac Event; Cardiac Implantable Electronic Device
MeSH Terms: conditions — Sleep Wake Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with low burden of sleep-disordered breathing
  Interventions: Diagnostic Test: Device interrogation
- Patients with high burden of sleep-disordered breathing
  Interventions: Diagnostic Test: Device interrogation

INTERVENTIONS:
Diagnostic Test: Device interrogation — All devices are interrogated at every follow-up, and two questionnaires are performed 2 years after enrollment.
  Other Names: Berlin Questionnaire; EuroQol five dimensions questionnaire

SUMMARY:
This prospective multicenter registry study aims to determine whether device-detected sleep-disordered breathing events are associated increased risk of cardiac arrhythmias or other cardiovascular outcomes.

DETAILED DESCRIPTION:
The prevalence of SDB high in patients with cardiac implantable electronic device (CIED). Recently, device-detected SDB events showed a correlation with sleep-disordered breathing (SDB) diagnosed by polysomnography. Thus, CIED will facilitate early detection and monitoring of SDB in patients with CIEDs. Few studies investigated prognostic value of CIED-detected SDB in risk of cardiovascular events. Therefore, the primary aim is to determine whether device-detected SDB are associated with increased risk of cardiac arrhythmias or other cardiovascular morbidities using a prospective multicenter registry.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 19years
* CHA2DS2VASc score ≥ 1 in male or ≥ 2 in female

Exclusion Criteria:

* CIED without atrial lead
* persistent or permanent atrial fibrillation (AF) or flutter
* history of catheter of surgical ablation of AF
* valvular steno-insufficiency more than moderate degree
* chronic obstructive pulmonary disease
* under current treatment for sleep-disordered breathing
* life expectancy < 1year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent implantation of cardiac implantable electronic device (CIED) with AP scan function (Boston Scientific.Inc) are eligible for the study during the first 3±1 months after CIED implantation.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with atrial fibrillation | from enrollment to last follow-up (2 years)
  cardiac implantable electronic device-detected or clinical atrial fibrillation

SECONDARY OUTCOMES:
Number of participants with complications associated with atrial fibrillation | from enrollment to last follow-up (2 years)
  thromboembolic events, heart failure, ablation therapy for atrial fibrillation
Number of participants with ventricular arrhythmia | from enrollment to last follow-up (2 years)
  cardiac implantable electronic device-detected or clinical ventricular arrhythmia

OTHER OUTCOMES:
Number of participants with major adverse composite events | from enrollment to last follow-up (2 years)
  cardiac death, stroke, atrial fibrillation or flutter, ventricular tachyarrhythmia, hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, PhD, Principal Investigator — Samsung Medical Center
Locations (15):
- South Korea (15):
  - Samsung Changwon Medical Center, Changwon
  - Chungbuk National University Hospital, Chungju
  - Chonnam National University Hospital, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Yeongnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Sejong General Hospital, Sejong
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gwag HB, Park Y, Lee SS, Kim JS, Park KM, On YK, Lee DI, Shin DG, Choi EK, Kang GH, Park HS, Park HW, Shim JM, Uhm JS, Kim J, Kim JH, Kang KW, Park SW, Oh YS, Cho Y, Lee YS, Park SJ. Rationale, design, and endpoints of the 'DEvice-Detected CArdiac Tachyarrhythmic Events and Sleep-disordered Breathing (DEDiCATES)' study: Prospective multicenter observational study of device-detected tachyarrhythmia and sleep-disordered breathing. Int J Cardiol. 2019 Apr 1;280:69-73. doi: 10.1016/j.ijcard.2019.01.045. Epub 2019 Jan 15. PMID 30665804